CLINICAL TRIAL: NCT00497380
Title: Arginine Feeding: a Novel Strategy to Improve Protein Metabolism in Cancer and the Response to Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 81167
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Protein Metabolism
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arginine enriched nutrition (Experimental)
  Interventions: Dietary Supplement: Arginine
- Nutrition (Placebo Comparator)
  Interventions: Dietary Supplement: Arginine

INTERVENTIONS:
Dietary Supplement: Arginine — Oral nutritional supplement

SUMMARY:
Muscle catabolism is a major problem in cancer patients undergoing surgery as it negatively affects post-operative recovery. Recent evidence exists that protein metabolic changes are already apparent in cancer before muscle wasting is being present. In line, patients with breast cancer, generally characterized by a normal nutritional status, were recently found to be arginine deficient. Arginine deficiency in cancer can be explained by: 1) Reduced arginine availability, due to exhaustion of endogenous (muscle) sources of arginine 2) Enhanced arginine catabolism, due to conversion of arginine by arginase, which is abundant in tumors. Protein is the most important endogenous source of arginine. Arginine deficiency will lead to a negative feedback loop in cachexia by promoting protein breakdown in an attempt to restore plasma arginine levels. We hypothesize that pre-operative arginine supplementation in breast cancer patients diminishes the occurrence of muscle wasting after surgery by 1) normalizing arginine availability pre-operatively, resulting in conservation of protein, 2) diminishing the catabolic effects of surgery by supplying exogenous arginine for the post-operative response, 3) enhancing the anabolic capacity to feeding through supplying substrate for protein synthesis.

DETAILED DESCRIPTION:
In the present proposal, the effects of surgery and cancer will be examined by comparing subjects undergoing breast surgery because of malignancy vs. prophylactic reasons (aim 1). Furthermore, the effects of one-week pre-operative protein feeding with or without enrichment with arginine on post-operative protein metabolism (aim 2) will be investigated in the cancer group. Variables of interest are: 1. Whole-body and skeletal muscle protein metabolism, whole body arginine turnover and de-novo arginine production rate, and the anabolic capacity to feeding(assessed by stable isotope methodology). 2. Body weight, muscle mass and functional status, score for well-being (assessed by Profile of Mood State and Mini Mental State).

In the present study, we propose that a nutritional supplement that is high in protein content and enhanced in arginine will be more effective than a typical commercial nutritional supplement in diminishing the catabolic effects of surgery in subjects with cancer, thereby optimizing their quality of life. If this is found to be the case, this would provide the basis for reformulating the nutritional composition in accord with the effects of cancer and surgery on protein metabolism.

ELIGIBILITY:
Inclusion Criteria:

Cancer groups (for aims 1 and 2)

1. Recently diagnosed (up to 4 weeks prior to treatment for cancer) with stage I, II or III invasive breast cancer
2. Undergoing mastectomy
3. Age greater than 30 years
4. Ability to sign informed consent
5. Good performance status defined by ECOG scale 0,1 or 2 (see CRF performance status)

Control group (for aim 1)

1. Age greater than 30 years
2. Undergoing prophylactic mastectomy
3. Ability to sign informed consent
4. Good performance status defined by ECOG scale 0,1 or 2 (see CRF performance status)

Exclusion Criteria:

All groups (aim 1 and 2)

1. Body weight loss of greater than 10% in the past 3 months
2. Previous anti-cancer therapy (e.g. chemotherapy or radiotherapy) or surgery less than 4 weeks prior to the experiment
3. Diagnosed diabetes type I or II
4. Untreated metabolic diseases including liver or renal disease
5. Any documented autoimmune disease
6. Use of corticosteroids, beta-antagonists or nitrovasodilators
7. Use of supplements enriched with amino acids
8. Presence of acute illness or metabolically unstable chronic illness
9. Unstable heart disease requiring therapy or recent myocardial infarction (less than 1 year)
10. Current alcohol or drug abuse (ETOH more than 2 servings per day)
11. Allergy/intolerance to any of the ingredients of the study products
12. Any other condition deemed by the PI and the study physician as exclusion or that interferes with proper conduct of the study/ safety of the patient.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08-18 (Actual); Primary Completion 2012-02-04 (Actual); Study Completion 2012-02-04 (Actual)

PRIMARY OUTCOMES:
Net protein balance | end of study

SECONDARY OUTCOMES:
Arginine turnover | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Deutz, M.D., Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Engelen MPKJ, Klimberg VS, Allasia A, Deutz NEP. Major surgery diminishes systemic arginine availability and suppresses nitric oxide response to feeding in patients with early stage breast cancer. Clin Nutr. 2018 Oct;37(5):1645-1653. doi: 10.1016/j.clnu.2017.07.019. Epub 2017 Aug 5. PMID 28826699